CLINICAL TRIAL: NCT04170556
Title: The GOING Study: Regorafenib Followed by Nivolumab in Patients With Hepatocellular Carcinoma Progressing Under Sorafenib or After Discontinuation of Atezolizumab Plus Bevacizumab
Brief Title: Regorafenib Followed by Nivolumab in Patients With Hepatocellular Carcinoma (GOING)
Acronym: GOING
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOING; 2019-003108-10 (EudraCT Number)
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular; sorafenib; regorafenib; nivolumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib; Nivolumab

STUDY DESIGN:
Intervention Model Description: Regorafenib followed by Nivolumab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib plus Nivolumab (Experimental): Regorafenib will be initiated at full dose (160 mg/day; 3 weeks on and 1 week off) in monotherapy for the first 8 weeks. After week 8, regorafenib will be continued in combination with nivolumab, until symptomatic tumor progression, unacceptable adverse events, patient decision or death
  Interventions: Drug: Regorafenib; Drug: Nivolumab

INTERVENTIONS:
Drug: Regorafenib — Regorafenib 160 mg/day 3 weeks on and 1 week off
Drug: Nivolumab — Nivolumab at the dose of 1.5 mg/kg, 3 mg/kg or 240 mg/infusion every 2 weeks. Dose will be adjusted depending on the incidence of adverse events

SUMMARY:
Regorafenib is an oral tumour deactivation agent that potently blocks multiple protein kinases, including kinases involved in tumour angiogenesis (VEGFR1, -2, -3, TIE2), oncogenesis (KIT, RET, RAF-1, BRAF, BRAFV600E), metastasis (VEGFR3, PDGFR, FGFR) and tumour immunity (CSF1R). In particular, regorafenib inhibits mutated KIT, a major oncogenic driver in gastrointestinal stromal tumours, and thereby blocks tumour cell proliferation.

Regorafenib has shown in clinical trials an acceptable benefit-risk across different tumor types, including colorectal cancer (CRC), GastroIntestinal Stromal Tumors (GIST) and HCC.

The most frequently observed adverse drug reactions (≥30%) in patients receiving regorafenib are pain, hand-foot skin reaction (HFSR), asthenia/fatigue, diarrhea, decreased appetite and food intake, hypertension, and infection.

Nivolumab is a human immunoglobulin G4 (IgG4) monoclonal antibody to the programmed death (PD)-1 receptor, blocking the interaction with PD-ligand (PD-L)1/PD-L213 and restoring T-cell-mediated antitumor activity. Nivolumab was evaluated in second-line the CheckMate 040 Study (Escalation and Expansion cohort.

In both cohorts of the CheckMate 040 Study, the safety profile was acceptable and there were no reported nivolumab-related deaths. In the dose-expansion cohorts from the Phase 1/2 CheckMate 040 Study, 65% of patients had treatment-related adverse events (TRAEs) of any grade 18% with Grade 3 or 4 TRAEs with fatigue, pruritus, and rash being the most common. Elevation of aspartate transaminase (AST) and alanine transaminase (ALT) were the most frequent Grade 3-4 TRAEs. AST/ALT elevations, however, were generally asymptomatic and readily managed.

For this reason, the rationale of this Phase I/IIa trial is to optimize the action of regorafenib and nivolumab but bearing in mind the potential impact of the drug-interaction and enhancement of the severity and/or frequency of adverse events. Thus, regorafenib will be administered as monotherapy during the first 2 cycles (each cycle is 3 weeks on plus 1 week off) of treatment to enhance T cell trafficking and infiltration into the tumor bed to increase the benefits of anti-PD-PD-L1, specific stimuli while emitting Damage-associated molecular patterns (DAMPs), followed by regorafenib plus nivolumab to impact step 7 of the cancer immunity cycle described by Chen.

The anti-PD-L1 effect under hypoxia was evaluated by Noman et al in a tumor model and they postulated that the abrogated myeloid-derived suppressor cells (MDSC)-mediated T cell suppression is achieved in part by modulating the cytokine production (IL-6 and IL-10). Specifically, hypoxia could promote immunosuppression by reducing the cytotoxic efficacy of immune cells, by increasing the peri-tumoral immunosuppressive cell populations infiltration of and priming the expression of immunosuppressive cytokines.

Current options for first line are sorafenib and atezolizumab-bevacizumab. Lenvatinib has been shown to be non-inferior to sorafenib, but it is less frequently used and its toxicity profile mandates a stringent selection of patients. Sorafenib shares some molecular targets with regorafenib, but this has specific action against VEGFR-2, VEGFR-3, Tie-2, PDGFR, FGFR-1, c-Kit, RET and p38-alpha7. Both are antiangiogenic as bevacizumab, but while bevacizumab is limited to the VEGF pathway, they act on several additional target involved in cancer progression. Atezolizumab and nivolumab target the PD1 checkpoint but acting at different levels: PD-1 receptor for Nivolumab and PD-L1 for Atezolizumab. This implies a difference and if resistance to one of the antibodies emerges during treatment, the use of the other one may overcome such key event leading to treatment failure. Recently, the combination of tremelimumab and durvalumab improved OS in comparison to sorafenib; in addition, durvalumab monotherapy was not inferior to sorafenib.

The aim of this study is to do a sequential treatment combining regorafenib, second- line treatment in hepatocellular carcinoma (HCC) with anti PD-1 to enhance the outcome of patients based on the synergy between both drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age or older.
2. Diagnosis of HCC based on histology or non-invasive criteria if the patients are cirrhotic according to AASLD guidelines.
3. Adequate liver function
4. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 to 1.
5. Adequate hematologic profile
6. Adequate renal function
7. All but sorafenib-related dermatologic adverse events must be grade I according to Common Terminology Criteria for Adverse Events (CTCAE) v.5.0. Early dermatologic adverse events related to first-line treatment must be resolved before starting regorafenib.
8. Patients with Hepatocellular Carcinoma

   * Who develop radiological tumor progression on sorafenib treatment within the 2 months of inclusion in the study and either:

     1. who are candidates to regorafenib treatment according to the definition in the RESORCE trial or
     2. who tolerated between 200 and 400 mg of sorafenib for at least 30 days and who did not experience adverse events of grade 3 or more (excluding dermatologic adverse events)(Cohort A).
   * After discontinuation of atezolizuamab in combination with bevacizumab because of tumor progression or treatment related toxicity (Cohort B). Note that patients should have received at least 2 doses of atezolizumab in combination with bevacizumab.
9. All subjects must have at least one measurable lesion by RECIST 1.1 criteria. Lesions previously treated by percutaneous ablation or TACE must not be considered as target lesion, only naïve target lesions.
10. Subjects may be non-infected or have active chronic HCV or HBV infection.
11. Subjects must consent to perform 2 hepatic or extra-hepatic tumor biopsies, the first one within 4 weeks before starting regorafenib (this biopsy should be performed at least 5-7 days after the last dose of sorafenib and 21 days after the last dose of atezolizumab in combination with bevacizumab) and the second-one before starting the combination phase (regorafenib plus nivolumab) of the study, allowing the acquisition of a tumor sample for performance of correlative studies.
12. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to the start of study drug.
13. Women must not be breastfeeding.
14. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug plus 90 days for a total of 31 weeks post-treatment completion
15. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements.
16. WOCBP must agree to follow instructions for method(s) of contraception from the time of enrollment for the duration of treatment with study drug plus 5 half-lives of study drug plus 30 days for a total of 23 weeks post treatment completion.

Exclusion Criteria:

1. Subjects with myocardial infarction in the last year or active ischemic heart disease
2. Subjects with any history of clinically meaningful variceal bleeding within the last three months.
3. Subjects with severe peripheral arterial disease
4. Subjects with cardiac arrhythmia under treatment with drugs different from beta-blockers or digoxin.
5. Subjects with clinically meaningful ascites defined as ascites requiring non-pharmacologic intervention within 6 months prior to the first scheduled dose.
6. Subjects with any history of encephalopathy within the last 12 months or requirement for medications to prevent or control encephalopathy.
7. Unfeasibility to fulfill the follow-up schedule
8. Co-infection with hepatitis B and C.
9. Prior malignancy active within the previous 3 years
10. Subjects with any active autoimmune disease or history of known or suspected autoimmune disease
11. Positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) defining opportunistic infection within the last year, or a current CD4 count < 350 cells/μL. Patients with HIV infection are eligible if :

    1. They do not have another active viral infection.
    2. They have received antiretroviral therapy (ART*) for at least 4 weeks prior to randomization, as clinically indicated.
    3. They continue on ART as clinically indicated while enrolled on study.
    4. CD4 counts and viral load are monitored per standard of care by a local health care provider.

    (*) The ART regimen includes drugs that are permitted according to protocol. An evaluation by the infectious disease specialist should be provided to the Medical Monitor (MM) prior to the enrollment.
12. Known active drug or alcohol abuse.
13. Prior therapy with an anti-PD-1, anti-PD-L1 (other than atezolizumab), anti-PD-L2, anti-CD137, or anti-Cytotoxic T-Lymphocyte Antigen 4 antibody (anti-CTLA-4 antibody)
14. Prior monotherapy treatment with any tyrosine kinase inhibitor in first line other than sorafenib.
15. Prior organ allograft or allogeneic bone marrow transplantation
16. All but dermatologic toxicities attributed to first-line treatment must have resolved to Grade 1 (NCI CTCAE version 5) or baseline before administration of study drug. Subjects with toxicities attributed to first-line treatment therapy that are not expected to resolve and result in long-lasting sequelae are not permitted. Neuropathy must have resolved to Grade 2 (NCI CTCAE version 5). Dermatologic toxicities must be resolved.
17. Active bacterial or fungal infections requiring systemic treatment within 7 days.
18. Use of other investigational drugs (drugs not marketed for any indication) within 28 days or at least 5 half-lives (whichever is longer) before study drug administration.
19. Known or underlying medical conditions that, in the Investigator's opinion, would make the administration of the study drug hazardous to the subjects or obscure the interpretation of toxicity determination or adverse events.
20. Subjects with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of study drug administration.
21. Laboratory evidence of any underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events
22. History of severe hypersensitivity reactions to other monoclonal antibodies or regorafenib.
23. History of allergy to study drug components.
24. WOCPB who are pregnant or breastfeeding.
25. Women with a positive pregnancy test at enrollment or prior to administration of study medication.
26. Prisoners or subjects who are involuntarily incarcerated.
27. Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness
28. Inability to comply with restrictions and prohibited activities/treatments.
29. Subjects in the Child-Pugh classes B≥7 points or C are not allowed to be recruited into this trial.
30. subjects with uncontrolled arterial hypertension.
31. Concomitant anticoagulation, at therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, low molecular weight heparin (LMWH), thrombin or coagulation factor X (FXa) inhibitors, or antiplatelet agents (eg, clopidogrel).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 24 months
  Rate of adverse events (AE)
Incidence of related Treatment-Emergent Adverse Events | Up to 24 months
  Rate of related-AEs
Incidence of Treatment-Emergent Adverse Events | Up to 24 months
  Rate of death

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 24 months
  Time from the date of start of treatment until the date of death
Time to progression (TTP) | Up to 24 months
  Time from the date of start of treatment until the date of objective disease progression or death
Objective response rate (ORR) | Up to 24 months
  Time from the date of start of treatment until the date of objective response
Pattern of progression | Up to 24 months
  Time from the date of start of treatment until the date of objective response
Post-progression survival (PPS) | Up to 24 months
  Time from the date of disease progression until the date of death
Rate of patients who develop new extra-hepatic spread | Up to 24 months
  Time from the date of start of treatment until the date of objective new extra-hepatic progression
Serum and tissue marker characterization | Up to 24 months
  Time from the date of start of treatment until the date of objective disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Maria Reig, MD, Principal Investigator — BCLC group. Liver Unit. Hospital Clinic. Ciberehd
Locations (7):
- Spain (7):
  - Hospital Clinic, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Gregorio Marañon, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Central de Asturias, Oviedo
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: Undecided